CLINICAL TRIAL: NCT05180682
Title: Effectiveness of Supervised Training Program on Mobility and Balance Confidence in Individual With Lower Limb Amputation: A Quasi-Experimental Study
Brief Title: Effectiveness of Supervised Training Program on Mobility and Balance Confidence in Individual With Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCS University System (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr. Hazrat Bilal PT, Principal Invistigator, Khyber Medical University Peshawar
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMU/IPMR/MS
Record Dates: First submitted 2021-12-19; First posted 2022-01-06 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Amputation
Keywords: Lower limb Amputation; Balance; Mobility

STUDY DESIGN:
Intervention Model Description: Participants were non randomly allocated to two groups and and were analyzed in the end of the study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised (Experimental): This group training was supervised by the health care provider.
  Interventions: Other: Gait Training
- Non-Supervised (Active Comparator): This group was non-supervised.
  Interventions: Other: Gait Training

INTERVENTIONS:
Other: Gait Training — the physical therapist will provide different protocol at different weeks in the following way.
  first week: first fitting and initial Gait training second week: Specific Gait Training third week: Advance Gait Training fourth week: Functional Training

SUMMARY:
It was quasi experimental study where the researchers assess the effectiveness of supervised training program on mobility and balance confidence in individual with lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 15-55 years.
2. Both genders: (male and females).
3. Trans-tibial amputation
4. Patients involved in prosthetic rehabilitation (strengthening, balance training, stretching exercises and gait training).

Exclusion Criteria:

1. Patient with cognitive problem.
2. Infection
3. Neuromas
4. Limb swelling

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Balance confidence | One month
  Balance was assessed through Activity-specific balance confidence. Its a 16-item questionnaire where patients' rate their confidence while doing activities.
  Scoring from 0-100 (0 is no confidence and 100 is full confidence) Paper survey, 5-10 mins for administration. No Training required.
Mobility | One month
  Mobility was assessed through loco-motor capabilities index. The loco-motor capabilities index is a disease-specific, self-administered instrument for assessing locomotor abilities generally considered essential for basic and advanced ADLs of people with lower-limb amputation and an enabling factor associated with long-term prosthetic use. It is easily administered and quickly completed.
  It is composed of 14 questions The LCI can be divided into two 7-item subscales that cover basic (items 1, 4, 5, 8-11) and advanced (items 2, 3, 6, 7,12-14) activities, respectively. Higher scores reflect greater locomotor capabilities with the prosthesis and less dependence on assistance. Maximum score = 56, Minimum score = 0

CONTACTS AND LOCATIONS:
Overall Officials: Hazrat Bilal, MSPT, Principal Investigator — Khyber Medical University Peshawar
Locations (1):
- Pakistan Institute of Prosthetic and Orthotic Sciences, Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No